CLINICAL TRIAL: NCT05422820
Title: The Argentina Brief Colonoscopy Difficulty Score (ABCD): A Novel Tool to Estimate the Technical Difficulty of Colonoscopy With Caecal Intubation
Brief Title: The Argentina Brief Colonoscopy Difficulty Score (ABCD)
Acronym: ABCD
Status: Completed | Type: Observational
Sponsor: Institute of Gastroenterology and Advance Endoscopy (Other)
Collaborators: Austral University, Argentina (Other); Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Principal Investigator, Manuel Valero, Principal investigator - Physician - GI Attending, Institute of Gastroenterology and Advance Endoscopy
Other Study IDs: IGEA01-2022
Record Dates: First submitted 2022-06-12; First posted 2022-06-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Diagnoses Disease; Polyp of Colon; Adenoma Colon
Keywords: Colonoscopy; Quality of health care; Endoscopist; Technical difficulty
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic high-definition white-light (HDWL) colonoscopy — All participants will undergo to colonoscopy examination performed by competent/junior or expert/senior endoscopists (>150-400 or >400 previous colonoscopies, respectively). Bowel preparation was performed using different solutions, according to the clinical discretion of the attending, who indicated colonoscopy. After deep sedation by intravenous propofol with or without fentanyl or midazolam administration, a water-assisted colonoscopy was performed using a high-definition (HD) scope with white light (WL). Colonoscope trademark differs among participant centres.

SUMMARY:
Colonoscopy completion by caecal intubation seldom represents a significant effort for the endoscopist. In this situation, additional techniques are necessary to achieve this goal: patients' manual abdominal compression, postural changes, and endoscopist relay. To date, no tool allows colonoscopy technical difficulty grading.

This study pursues to describe the frequency of additional techniques for caecal intubation in a large sample of Argentinians in different centres who undergo colonoscopy for attending purposes, to develop a novel score for assessing colonoscopy technical difficulty.

DETAILED DESCRIPTION:
Colonoscopy is the most performed digestive endoscopy procedure worldwide. It is indicated for colorectal cancer screening, pre-existence surveillance, diagnostic approach in symptomatic patients, and therapeutic purposes. Bowel preparation is the most crucial quality criterion that guarantees appropriate colonic mucosa assessment. Other colonoscopy quality criteria included a colonoscope withdrawal time above 6 to 10 minutes and colonoscopy completion by caecal intubation.

Besides bowel preparation, some situations limit caecal intubation: stenosis, diverticulitis, or haemodynamic instability. In the absence of one of those situations or similar, caecal intubation must be the goal to be achieved by every endoscopist. However, it sometimes represents a significant effort for the endoscopist. It can require additional techniques such as manual abdominal compression, postural changes, colonoscopy restart, and another endoscopist's new attempt. Also, this increases caecal intubation time by over 10 minutes, more anaesthesia and post-colonoscopy abdominal pain, with a higher risk of unnoticed lesions.

To the best of our knowledge, there is no standard definition for colonoscopy technical difficulty in terms of caecal intubation or any tool that grades it based on previously mentioned additional techniques. For the moment, developed tools such as the Difficult Colonoscopy Score (DCS) to consider patients' pre-colonoscopy factors such as age, body mass index (BMI), sleep quality, and endoscopist experience. Other tools are based on a qualitative appreciation of the technical difficulty.

A tool that documents those endpoints constitutes an additional objective quality criterion for colonic mucosa assessment, with critical change management during intra-colonoscopy and post-colonoscopy. Noticed a technically difficult colonoscopy deserves a more prolonged withdrawal time, more photo documentation, a more cautious discharge, more detailed patient instructions, and a personalised follow-up directed to adverse events warnings. A patient with a previous technically difficult colonoscopy will be planned for an earlier next colonoscopy, with a risk assessment independently on the age, pre-colonoscopy consulting with detailing of more potential adverse events, planned in a particular time and with a different anaesthesia planning, and even performed by a more experienced endoscopist or in a referral centre.

This study pursues to describe the frequency of additional techniques for caecal intubation in a large sample of Argentinians in different centres who undergo colonoscopy for attending purposes, to develop a novel score for assessing colonoscopy technical difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colonoscopy indication due to colorectal cancer screening, pre-existence surveillance, or diagnostic approach in symptomatic patients.
* Patients with colonoscopy indication due to therapeutic purposes, but with the intention of caecal intubation.

Exclusion Criteria:

* Patients with a previous colonoscopy performed by the attending centre in the last three months.
* Patients with a Boston Bowel Preparation Score (BBPS) ≤1 in at least one colon segment (ascending, transverse, descending).
* Patients with any situations which does not allow caecal intubation: colorectal stenosis, diverticulitis, the indication of proctosigmoidoscopy for assessing ulcerative colitis, or intraprocedural haemodynamic instability, among others.
* Patients with any contraindication for an invasive procedure: uncontrolled coagulopathy, kidney/liver failure or any comorbidity with an important impact on cardiac risk assessment or physical status: New York Heart Association (NYHA) risk III/IV, or American Society Association (ASA) risk III-V, respectively.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication of colonoscopy with caecal intubation, regardless of clinical purpose.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Argentina Bowel Complexity and Colonoscopy technical Difficulty score (ABCD) | Six months
  Per each colonoscopy, there were documented:
  1. The number of cases in which caecal intubation (CI) was or was not achieved.
  2. Number of endoscopists who participated until caecal intubation, with the respective learning curve experience (expert/senior vs. non-expert/junior);
  3. Requirement of restart colonoscopy (regardless of the responsible endoscopist);
  4. Requirement of at least one postural change (from lateral to supine or vice versa);
  5. Requirement of manual abdominal pressure.
  ABCD score ranges from 0 to IV:
  0: no difficulty. I: low difficulty. CI was issued after an effective abdominal compression. II: mild difficulty. CI was issued after a partial effective abdominal compression.
  III: high difficulty. CI was issued after body rotation or change of endoscopist.
  IV: very high difficulty. Declined cecal intubation after several attempts using additional techniques.

SECONDARY OUTCOMES:
Caecal intubation and colonoscope withdrawal time | During procedure: no more than 30 minutes.
  The caecal intubation time (CIT) is the time (mm:ss) from colonoscope insertion to the anal margin until caecal intubation (or its desertion after several attempts). Biopsy or therapeutic time will not be considered for this research.
  The colonoscope withdrawal time (CWT) is the time (mm:ss) from caecal intubation (or its desertion after several attempts) until the returning to the anal margin after assessing the colonic mucosa thoroughly. Biopsy or therapeutic time will not be considered for this research.
Required anaesthesia dose | During procedure: no more than 30 minutes.
  Dose of propofol (mg) with or without fentanyl (mcg) or midazolam (mg) used during colonoscopy, following anaesthesia record.
Post-colonoscopy pain | Six months
  Level of pain described by the patient one-hour post-colonoscopy. A general practitioner blind to the ABCD findings will ask the patient about pain from 1 (one) to 10 (ten), showing the Wong-Baker face pain rating scale, a type of visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel Valero, Bahía Blanca, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia H, Wang L, Luo H, Yao S, Wang X, Zhang L, Huang R, Liu Z, Kang X, Pan Y, Guo X. Difficult colonoscopy score identifies the difficult patients undergoing unsedated colonoscopy. BMC Gastroenterol. 2015 Apr 9;15:46. doi: 10.1186/s12876-015-0273-7. PMID 25886845
- [Background] Fritz CDL, Smith ZL, Elsner J, Hollander T, Early D, Kushnir V. Prolonged Cecal Insertion Time Is Not Associated with Decreased Adenoma Detection When a Longer Withdrawal Time Is Achieved. Dig Dis Sci. 2018 Nov;63(11):3120-3125. doi: 10.1007/s10620-018-5100-x. Epub 2018 May 3. PMID 29721773
- [Background] Allen JI. Quality measures for colonoscopy: where should we be in 2015? Curr Gastroenterol Rep. 2015 Mar;17(3):10. doi: 10.1007/s11894-015-0432-6. PMID 25740247
- [Background] ASGE Technology Committee; Trindade AJ, Lichtenstein DR, Aslanian HR, Bhutani MS, Goodman A, Melson J, Navaneethan U, Pannala R, Parsi MA, Sethi A, Sullivan S, Thosani N, Trikudanathan G, Watson RR, Maple JT. Devices and methods to improve colonoscopy completion (with videos). Gastrointest Endosc. 2018 Mar;87(3):625-634. doi: 10.1016/j.gie.2017.12.011. No abstract available. PMID 29454445
- [Background] Clancy C, Burke JP, Chang KH, Coffey JC. The effect of hysterectomy on colonoscopy completion: a systematic review and meta-analysis. Dis Colon Rectum. 2014 Nov;57(11):1317-23. doi: 10.1097/DCR.0000000000000223. PMID 25285700